CLINICAL TRIAL: NCT06456125
Title: Safety and Efficacy Of Amber Peripheral Liquid Embolic System: a First-in-HumAn & PivotaL Study
Brief Title: Safety and Efficacy Of Amber Peripheral Liquid Embolic System
Acronym: OPAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LVD Biotech S.L (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: amber SEL-P-01
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Vascular Anomalies; Hemorrhage; Aneurysm; Pseudoaneurysm; Varicose Veins; Portal Vein Embolization; Hypervascular Tumor; Type II Endoleak; Pathological Organ
Keywords: liquid embolic agent; peripheral vascular embolization; embolization; endovascular therapy; interventional radiology
MeSH Terms: conditions — Vascular Malformations; Hemorrhage; Aneurysm; Aneurysm, False; Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amber SEL-P Treatment (Experimental): Patients requiring peripheral embolization: vascular anomalies, hemorrhages, aneurysms, and pseudoaneurysms, varicose veins (including varicocele and pelvic congestion syndrome), portal vein, hypervascular tumors, type -II endoleaks, and pathological organs.
  Interventions: Device: amber SEL-P Peripheral Liquid Embolic System

INTERVENTIONS:
Device: amber SEL-P Peripheral Liquid Embolic System — Transcatheter arterial or venous embolization with the liquid embolic agent amber SEL-P embolization across seven different indications for peripheral embolization.

SUMMARY:
A prospective, single-arm, multicenter, open-label, First-in-Human & Pivotal Study to assess the safety and efficacy of amber SEL-P in 70 patients requiring peripheral embolization: vascular anomalies, hemorrhages, aneurysms, and pseudoaneurysms, varicose veins, portal vein, hypervascular tumors, type -II endoleaks, and pathological organs.

The study will be divided into two consecutive stages. Stage I will be dedicated to testing the device's safety, followed immediately by stage II, aimed to test the device's efficacy. The overall study sample will be used to assess the device safety and efficacy in all the enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 and < 95 years presenting with one of the following indications:

  * Varicose vein embolization:

    * Pelvic congestion syndrome (uterine venous engorgement, and/or moderate or severe engorgement of the ovarian plexus, and/or filling of the veins across the midline or filling of vulvar or thigh varicosities, and/or reflux throughout the entire course of the ovarian vein.
    * Varicocele (symptomatic varicocele, and/or infertility or subfertility).
    * Varicose veins in patients with portal hypertension undergoing Transjugular Intrahepatic Portosystemic Shunt (TIPS) that require embolization.
  * Type II endoleak: Persistent type II endoleak and/or an associated sac expansion > 5 mm after 6 months or 10 mm after 12 months.
  * Insufficient liver remnant requiring portal vein embolization (PVE) before liver resection: Predicted insufficient liver remnant after surgery (≤20% in a normal liver, ≤30% in liver with intermediate disease without cirrhosis, and ≤40% in liver with cirrhosis)
  * Active arterial hemorrhage and/or pseudoaneurysm: Uncontrolled massive hemorrhage caused by tumor, trauma or arteriovenous shunt formation (congenital or acquired), and/or up to 3 bleeding sites in the same organ or anatomic region
  * Pathologic organ (i.e. non-functioning transplanted kidney, preoperative hip replacement, hypersplenism conditioning low platelet count; excluding brain)
  * Hypervascular tumors
  * Vascular anomalies

Exclusion Criteria:

* Patients with known hypersensitivity or allergy to amber-20, dimethylsulfoxide (DMSO) solvent, or contrast agent
* Previously failed embolization procedure, except for those treated with coils
* Patient in whom according to the investigator criteria a complete vascular occlusion would not be feasible in a single procedure
* Any condition that exposes the patient to a high risk for complications according to the investigator's criteria (e.g., but not limited to, non-correctable coagulopathy, uncontrolled sepsis, underlying life-threatening condition, etc.)
* Patients participating in another interventional study that has not completed it primary endpoint assessment.
* Pregnant or breastfeeding women.
* Patients unable or unwilling to provide a written informed consent.
* Recurrent varicose vein embolization
* Type II endoleak: with high flow or reflux that cannot be prevented using coils or balloon microcatheter, and high risk of medullar ischemic damage
* Active arterial bleeding and/or pseudo aneurysm with: severe hemodynamical instability (e.g., but not limited to, sustained hypotension [mean arterial pressure < 60 mmHg], tachycardia >120 beats/minute, requirement of high doses of vasopressors, etc.) at the moment of the procedure, and/or hb < 8 g/dL before the procedure, and/or retroperitoneal hemorrhages or hemoptysis, identification of spinal or medullar vessels.
* Central nervous system and central circulatory system vascular anomalies.
* Iodine contrast allergy

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peri-procedure serious adverse events related to amber SEL-P (Stage I) | Up to 24 hours after embolization procedure
  Rate of peri-procedure serious adverse events related to amber SEL-P (device-related but not related to the procedure) at 24 hours, adjudicated by an independent clinical events committee.
Rate of complete vascular occlusion (Stage II) | Embolization procedure day
  Rate of complete vascular occlusion as defined by angiography at the end of the procedure.

SECONDARY OUTCOMES:
Rate of any peri-procedure adverse events related to amber SEL-P (Stage I) | Up to 24 hours after embolization procedure
  Rate of any peri-procedure adverse events related to amber SEL-P (device-related but not related to the procedure) at 24 hours, adjudicated by an independent clinical events committee.
Rate of complete vascular occlusion according clinical indication (Stage II) | Embolization procedure day
  Rate of complete vascular occlusion as defined by angiography at the end of the procedure according to clinical indication.
  * Vascular anomalies (excluding the central nervous system and central circulatory system).
  * Hemorrhages, aneurysms, and pseudoaneurysms.
  * Varicose veins (including hemorrhoids, varicocele, and pelvic congestion syndrome).
  * Portal embolization.
  * Hypervascular tumors.
  * Type II endoleaks.
  * Pathological organs (renal grafts, hypersplenism).
Rate of peri-procedure serious adverse events related to amber SEL-P (Stage II) | Up to 24 hours after embolization procedure
  Rate of peri-procedure serious adverse events related to amber SEL-P (device-related but not related to the procedure) at 24 hours, adjudicated by an independent clinical events committee.

OTHER OUTCOMES:
Peri-procedure serious adverse event (Stage I and Stage II) | Up to 24 hours after embolization procedure
  Rate of peri-procedure serious adverse events related to amber SEL-P (device-related but not related to the procedure) at 24 hours, adjudicated by an independent clinical events committee.
Technical success (Stage I and Stage II) | Embolization procedure day
  Rate of complete vascular occlusion as defined by angiography at the end of the procedure
Peri-procedure adverse events (Stage I and Stage II) | Up to 24 hours after embolization procedure
  ate of any peri-procedure adverse events related to amber SEL-P (device-related but not related to the procedure) at 24 hours, adjudicated by an independent clinical events committee.
Technical success per indication (Stage I and Stage II) | Embolization procedure day
  Rate of complete vascular occlusion as defined by angiography at the end of the procedure according to clinical indication
Any Serious Adverse Events (Stage I and Stage II) | up to 6 moonths
  Total number of any serious adverse events
Any Adverse Events (Stage I and Stage II) | up to 6 moonths
  otal number of any adverse events
Survival rate (Stage I and Stage II) | up to 6 moonths
  Survival rate
Visual Analog Scale (VAS) injection (Stage I and Stage II) | Embolization procedure day
  Visual Analog Scale (VAS) to evaluate the pain at device injection (between 0: no pain to 10: intolerable pain)
Visual Analog Scale (VAS) varicose vein (Stage I and Stage II) | up to 6 moonths
  Visual Analog Scale (VAS) to evaluate pain improvement in patients with painful varicose vein embolization
Unanticipated uses of another liquid agent (Stage I and Stage II) | Embolization procedure day
  Total number of unanticipated uses of another liquid agent for embolization
Volume of amber SEL-P (Stage I and Stage II) | Embolization procedure day
  Mean volume of amber SEL-P used during the index procedure
Vials per patient of amber SEL-P (Stage I and Stage II) | Embolization procedure day
  Mean vials per patient of amber SEL-P used during the index procedure
Degree of occlusion (Stage I and Stage II) | Embolization procedure day
  Mean degree of occlusion of the target vessel(s).
Re-interventions (Stage I and Stage II) | up to 6 moonths
  Total number of re-interventions for the study procedure.
Clinical success | up to 6 moonths, depending on indication
  oVaricose vein embolization: absence of reflux on ultrasound Doppler at 1M FU, reduction in macroscopic varicose veins and or improvement of pain at least 2 points measured by means of visual analogue scale (VAS).
  oType II endoleaks: stability or reduction of the aneurysm's anteroposterior and transverse maximal diameters on a computed tomography (CT) scan at 6 months compared with baseline (4-mm growth threshold).
  oPVE: growth of the future liver remnant (FLR) by >15% assessed on a presurgical CT scan compared with baseline.
  oHemorrhage, aneurysm, pseudoaneurysm, pathologic organ: complete occlusion of the target vessel as assessed by angiography during the index procedure.
  o Hypervascular tumor and vascular anomalies : Correct devascularization of the treated lesion (intentionally complete or incomplete defined at the end of the procedure).
EQ-5D (Stage I and Stage II) | up to 6 moonths
  Baseline and follow-up patient's quality of life EQ-5D (unabbreviated: EuroQol 5-dimensions ). Health state index scores generally range from 0 (dead) to 1 (perfect health), with higher scores indicating higher health utility.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Gómez, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital Universitario Y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No